CLINICAL TRIAL: NCT04660552
Title: Transcranial Photobiomodulation for Reducing Autism Symptoms in Children
Acronym: TPBMASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JelikaLite LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19751975
Record Dates: First submitted 2020-11-16; First posted 2020-12-09 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-03

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: This is a Randomized, Placebo-controlled, Double Blind, Mixed Design study
Who Masked: Participant, Care Provider, Investigator
Masking Description: To minimize the bias, Jelikalight hired an independent pediatric psychiatrist, to act as a PI and supervise the study. The PI is blind (and will remain blind until the end of the study data collection and analysis) to the participants' condition. He will supervise data collection and analysis. The PI will supervise parental interviews. The PI will conduct before and after treatment testing of participants with CARS2. The PI will supervise analysis for raw data. Experimental and control groups will undergo the same experience apart from having the device turned on or turned off during the sessions. The participants (and their parents) will remain blind to their experimental condition, therefore, ensuring double blindness.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- CognilumTM (Experimental): During the study participants will be wearing the photobiomodulation device Cognilum. The device will administer the stimulation of near infrared light (830nm) to specific areas of the child's brain.
  Interventions: Device: Cognilum TM: Light Treatment Condition
- Placebo condition (Placebo Comparator): During the study participants will be wearing the photobiomodulation device. The device will not be turned on and therefore no brain stimulation with near infrared light (830nm) will be provided.
  Interventions: Device: Cognilum TM: Light Treatment Condition

INTERVENTIONS:
Device: Cognilum TM: Light Treatment Condition — The children will wear the CognilumTM device for up to 15 minutes at a time, twice a week, for a period of 8 weeks.

SUMMARY:
The hypothesis of the study is that photobiomodulation reduces symptoms of autism. Participants will be children between the ages of 2 and 6, who have been diagnosed with moderate to severe autism. Transcranial photobiomodulation will be administered to the children in the experimental condition twice a week for 8 weeks. Results will be measured through parental interviews, standardized CARS2 (Childhood Autism Rating Scales, 2nd Edition) and data collected from EEG.

DETAILED DESCRIPTION:
The CognilumTM System is a non-invasive device that uses infrared light (IR), delivered through light emitting diodes (LEDs) built into a head band worn by the patient during treatment.

The proposed clinical investigation is determined by the FDA to be a nonsignificant risk (NSR) device study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants between 2 years and 6 years of age (inclusive), of all races.
2. Previously diagnosed with moderate or severe ASD by a licensed professional.
3. Participants may be receiving any behavioral intervention therapy (e.g., ABA, Floor Time) during the course of the treatment. The final statistical analysis will control for the participants receiving behavioral therapies in control and experimental conditions. We expect the majority of the participants in both control and experimental conditions to be receiving behavioral therapies. There is no known interactions or complications of tPBM with behavioral therapy.
4. Parents of participants must understand the nature of the study.
5. Parents of participants must sign an IRB- approved informed consent form before initiation of any study procedures.
6. Parents of participants must have a level of understanding sufficient to communicate with the investigator and study coordinator, and to cooperate with all tests and examinations required by the protocol.
7. Participant child experiencing a major psychiatric disorder will be allowed to participate in the study provided they do not meet any exclusionary criteria.
8. The participant child is willing to participate in this study.

Exclusion Criteria:

1. Participant child is experiencing severe self-injurious behavior or severe aggressive behavior to self or others (within past 7 days).
2. Participant has been diagnosed with another psychiatric or neurological disorder (e.g. epilepsy) or have exhibited symptoms of major psychiatric disorders within the last 30 days.
3. Participant has an unstable medical condition (that requires clinical attention).
4. Participant has a significant skin condition at the procedure sites (i.e., hemangioma, scleroderma, psoriasis, rash, open wound or tattoo).
5. Participant has an implant of any kind in the head (e.g. stent, clipped aneurysm, embolised AVM, implantable shunt - Hakim valve).
6. Participant has receiving medication on a regular basis for Autism or any other medical condition.
7. Any use of light-activated drugs (photodynamic therapy) within 14 days prior to study enrollment (in US: Visudine (verteporfin) - for age related macular degeneration; Aminolevulinic Acid- for actinic keratoses; Photofrin (porfimer sodium) - for esophageal cancer, non-small cell lung cancer; Levulan Kerastick (aminolevulinic acid HCl) - for actinic keratosis; 5-aminolevulinic acid (ALA)- for non-melanoma skin cancer).
8. Current treatment with a psychotropic medication.
9. Investigator and his/her immediate family, defined as the investigator's child or grandchild.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuli Fradkin, MD, Principal Investigator — RDT Group NJ
Locations (2):
- United States (2):
  - Dr. Steingold Psychology PC, Brooklyn, New York
  - Dr. Steingold Psychology PC, New York, New York

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be available to other researchers

REFERENCES:
- [Background] Bosl WJ, Tager-Flusberg H, Nelson CA. EEG Analytics for Early Detection of Autism Spectrum Disorder: A data-driven approach. Sci Rep. 2018 May 1;8(1):6828. doi: 10.1038/s41598-018-24318-x. PMID 29717196
- [Background] Hamblin MR. Shining light on the head: Photobiomodulation for brain disorders. BBA Clin. 2016 Oct 1;6:113-124. doi: 10.1016/j.bbacli.2016.09.002. eCollection 2016 Dec. PMID 27752476
- [Background] Henderson TA, Morries LD. Near-infrared photonic energy penetration: can infrared phototherapy effectively reach the human brain? Neuropsychiatr Dis Treat. 2015 Aug 21;11:2191-208. doi: 10.2147/NDT.S78182. eCollection 2015. PMID 26346298
- [Background] Khuman J, Zhang J, Park J, Carroll JD, Donahue C, Whalen MJ. Low-level laser light therapy improves cognitive deficits and inhibits microglial activation after controlled cortical impact in mice. J Neurotrauma. 2012 Jan 20;29(2):408-17. doi: 10.1089/neu.2010.1745. Epub 2011 Sep 21. PMID 21851183
- [Background] Leisman G, Machado C, Machado Y, Chinchilla-Acosta M. Effects of Low-Level Laser Therapy in Autism Spectrum Disorder. Adv Exp Med Biol. 2018;1116:111-130. doi: 10.1007/5584_2018_234. PMID 29956199
- [Background] Weissman JR, Kelley RI, Bauman ML, Cohen BH, Murray KF, Mitchell RL, Kern RL, Natowicz MR. Mitochondrial disease in autism spectrum disorder patients: a cohort analysis. PLoS One. 2008;3(11):e3815. doi: 10.1371/journal.pone.0003815. Epub 2008 Nov 26. PMID 19043581
- [Result] Fradkin Y, De Taboada L, Naeser M, Saltmarche A, Snyder W, Steingold E. Transcranial photobiomodulation in children aged 2-6 years: a randomized sham-controlled clinical trial assessing safety, efficacy, and impact on autism spectrum disorder symptoms and brain electrophysiology. Front Neurol. 2024 Apr 26;15:1221193. doi: 10.3389/fneur.2024.1221193. eCollection 2024. PMID 38737349
- [Derived] Fradkin Y, Anguera JA, Simon AJ, De Taboada L, Steingold E. Transcranial photobiomodulation for reducing symptoms of autism spectrum disorder and modulating brain electrophysiology in children aged 2-7: an open label study. Front Child Adolesc Psychiatry. 2025 Jan 29;4:1477839. doi: 10.3389/frcha.2025.1477839. eCollection 2025. PMID 39944746

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CognilumTM | Placebo Condition
Started | 19 | 15
Completed | 16 | 14
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CognilumTM | Placebo Condition | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.9 (1.25) | 4.6 (1.16) | 4.6 (1.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 14 | 10 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 15 | 14 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 11 | 11 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Childhood Autism Rating Scales, Second Edition (CARS, 2nd Edition) [Mean (Standard Deviation); unit: units on a scale] — Childhood Autism Rating Scales, Second Edition (CARS, 2nd Edition), patients were evaluated at baseline, before any treatment was administered.
  CARS is a validated clinical rating scale that can be used by a trained clinician to rate items indicative of ASD after direct observation of the child.
  The scale consists of fifteen items that correspond to the different core domains (e.g., verbal communication, emotional response, and relationships with people) that can be affected by ASD.
  Total score (sum of all 15 sub-scales) can range from a low of 15 (no ASD) to a high of 60 (severe ASD).
  units on a scale | 43.5 (5.7) | 40.6 (7.2) | 43.5 (6.46)

OUTCOME MEASURES:

1. Primary Outcome: Change in Autism Symptoms
Description: Childhood Autism Rating Scales, Second Edition (CARS, 2nd Edition), patients were evaluated after conclusion of the study.
  CARS is a validated clinical rating scale that can be used by a trained clinician to rate items indicative of ASD after direct observation of the child.
  The scale consists of fifteen items that correspond to the different core domains (e.g., verbal communication, emotional response, and relationships with people) that can be affected by ASD.
  Total score (sum of all 15 sub-scales) can range from a low of 15 (no ASD) to a high of 60 (severe ASD).
  For the outcome measure we took the difference between the CARS score at the completion of the study and the CARS score at baseline.
Time Frame: 8 weeks
Population: The study enrolled children of both sexes aged two to six years, who had previously been diagnosed with ASD by a licensed professional according to the Diagnostic Statistical Manual of Mental Disorders, Fifth Edition (DSM V).
  Every participant was assessed using Childhood Autism Rating Scales, Second Edition (CARS, 2nd Edition).
  Participants were evaluated before the course of treatment (baseline) and after the course of treatment. Treatment duration was 8 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CognilumTM | Placebo Condition
Number analyzed (Participants) | 16 | 14
score on a scale | -9.87 (4.19) | -2.64 (7.99)
Statistical Analysis 1: Comparison: CognilumTM vs Placebo Condition; Test type: Equivalence — The post treatment cars scores of active and sham group will be statistically different as measured by independent sample t-test with p<.05; p = 0.01, t-test, 2 sided; Mean Difference (Net) = 7.23, 95% CI 2-sided [2.357 to 12.107], Standard Deviation 4.2

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | CognilumTM | Placebo Condition
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT04660552/Prot_003.pdf
  • Statistical Analysis Plan (2024-03-19): https://cdn.clinicaltrials.gov/large-docs/52/NCT04660552/SAP_004.pdf
  • Informed Consent Form (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT04660552/ICF_006.pdf